CLINICAL TRIAL: NCT04608578
Title: Evaluation of a Serious Game Aimed at Improving Mental Health in Youth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BC - 07288
Record Dates: First submitted 2020-10-24; First posted 2020-10-29 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Mental Health
Keywords: Suicide Prevention; Universal Suicide Prevention; Serious Game
MeSH Terms: conditions — Psychological Well-Being; Suicide Prevention | interventions — Silver

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group gain access to the game after filling in the baseline online questionnaire. The participants are asked to play at least two characters in the game. They have two weeks to play the game.
  Interventions: Behavioral: Silver
- Control group (No Intervention): Waitlist control group

INTERVENTIONS:
Behavioral: Silver — A serious game to improve mental health in youth
  Arms: Intervention group

SUMMARY:
The main goal of this study is to evaluate the effectiveness of a serious game aimed at improving mental health in teenagers aged 12-16 years old. This will test the effectiveness by studying the effect on emotion regulation strategies, coping strategies, the presence of cognitive errors and suicidal ideation. Participants will also be asked to evaluate the game. The study is a cluster-randomized controlled trial conducted in secondary schools in Flanders.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking
* having access to a smartphone or tablet

Exclusion Criteria:

* not being part of the selected classes in the participating schools

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
The Dutch version of the Questionnaire for the assessment of emotion regulation in children and adolescents (FEEL-KJ) | Baseline and posttest (after 2 weeks)
  A 90-item self-report instrument measuring seven adaptive, five maladaptive, and three external emotion (sadness, anger, and anxiety) regulation strategies. Each item is rated on a 5-point Likert scale from 1 = almost never to 5 = almost always. The score on the adaptive (ranging from 42-210), maladaptive (ranging from 30-150) and external (ranging from 18-90) subscales are considered. The higher the score on a subscale, the greater the disposition to cope with negative emotions in a certain way.

SECONDARY OUTCOMES:
Children's Coping Strategies Checklist -Revision 1 (CCSC-R1) | Baseline and posttest (after 2 weeks)
  3 subscales on cognitive coping strategies (i.e., optimism, control, and seeking understanding) are used. Each subscale has 4 items and all items are scored on a 4-point Likert scale from 1 = never to 4 = most of the time. For each subscale the minimum total score is 4 and the maximum score 16. The higher the mean score on the subscale, the more often the cognitive coping strategy is used.
Children's Negative Cognitive Error Questionnaire-Revised (CNCEQ-R) | Baseline and posttest (after 2 weeks)
  The scale assess cognitive Errors and has 5 subscales and 16 items in total. The items are rated on a 5-point Likert scale from 1 = not at all like I would think to 5 = almost exactly like I would think. Total scores range from 16-80. Higher scores reflect more distorted cognitive processes.
2 subscales of the EMO-check kids | Baseline and posttest (after 2 weeks)
  Two subscales of the EMO-Check kids are used i.e., Emotional clearness and Understanding emotions. They measure strategies to cope with emotions on a 5-point Likert scale from 0 = not at all to 4 = (almost) always. The score on a subscale ranges from 0 to 12. Higher score indicate more use a certain emotion regulation strategy.
Children's Depression Inventory, version 2 (CDI-2) | Baseline and posttest (after 2 weeks)
  A 28-item self-report scale measuring depressive symptoms experienced over the previous 2 weeks. Items are score on a scale from 0 to 2. Total scores range from 0 to 56. Higher scores indicate greater severity of depressive symptomatology.

OTHER OUTCOMES:
Game Evaluation | Posttest (after 2 weeks)
  14 statements regarding the effect, content and usefulness of the game. Items were rated on a 5-point Likert scale (1 = 'completely disagree'; 5 = 'completely agree').

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (14):
- Belgium (14):
  - De!Kunsthumaniora, Antwerp
  - KA Beveren, Beveren
  - VTI Brugge, Bruges
  - GO! Atheneum Denderleeuw, Denderleeuw
  - Kunsthumaniora Sint-Lucas, Ghent
  - Humaniora Kindsheid Jesu, Hasselt
  - Middenschool Kindsheid Jesu, Hasselt
  - GO! Atheneum Heist, Heist-op-den-Berg
  - RHIZO Hotelschool, Kortrijk
  - RHIZO Lyceum OLV Vlaanderen, Kortrijk
  - GO! Campus Redingenhof Leuven, Leuven
  - GO! Atheneum Ninove, Ninove
  - De Burgerschool, Roeselare
  - PITO Stabroek, Stabroek

IPD SHARING:
Plan to Share IPD: No